CLINICAL TRIAL: NCT05708183
Title: Healthy Mums, Healthy Babies in Ethiopia: a Cluster-randomized Trial to Evaluate the Programme Effectiveness of a Multiple Micronutrient Supplement Delivered to Pregnant Women Through Routine Antenatal Care to Improve Newborn Birthweight
Brief Title: Healthy Mums, Healthy Babies: Multiple Micronutrient Supplementation in Ethiopia
Status: Recruiting | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Ethiopian Public Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: 101534IC
Record Dates: First submitted 2022-09-21; First posted 2023-02-01 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Birth Weight
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Districts that have substituted MMS for IFA as part of routine antenatal care
  Interventions: Dietary Supplement: Multiple micronutrient supplementation (MMS)
- Comparison: Districts that continue to deliver IFA as part of routine antenatal care
  Interventions: Dietary Supplement: Iron folate supplementation (IFA)

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient supplementation (MMS) — Ethiopia will distribute the UNIMMAP (United Nations International Multiple Micronutrient Antenatal Preparation) formulation that includes 30mg iron. The supplement contains 15 essential vitamins and minerals including: Retinol (Vitamin A-acetate) 800 μg; Vitamin E (as vitamin E-acetate) 10 mg; Vitamin D (as Cholecalciferol) 200 IU; Vitamin B1 (Thiamine mononitrate) 1.4 mg; Vitamin B2 (As Riboflavin) 1.4 mg; Vitamin B3 (As Nicotinamide) 18 mg; Vitamin B6 (as Pyridoxine 1.9 mg; Vitamin B12 (as Cyanocobalamin) 2.6 mg; Folic Acid 400 μg; Vitamin C (As Ascorbic Acid) 70 mg; Iron (As ferrous sulphate) 30 mg; Zinc (As zinc sulphate) 15 mg; Copper (as Copper Sulphate) 2 mg; Selenium (as Sodium selenite) 65 μg; Iodine (as Potassium Iodate) 150 μg.
  Groups: Intervention
Dietary Supplement: Iron folate supplementation (IFA) — IFA delivered as part of routine antenatal care, according to current policy
  Groups: Comparison

SUMMARY:
Background: This programme effectiveness study responds to the need for evidence on the effect on birthweight of switching from iron-folic acid supplementation (IFA) to multiple micronutrient supplementation (MMS) as part of routine antenatal care in Ethiopia. A 2019 meta-analysis of trial data reported a mean improvement of 35g in newborn birthweight amongst newborns born to women who took MMS in pregnancy compared to those who took IFA. Responding to this evidence, in 2020 the World Health Organisation updated its global guideline on MMS from 'not recommended' to 'recommended in the context of rigorous research'. The guideline identifies priority research being 'to establish the impact of switching routine antenatal IFA to MMS on important health outcomes, equity, acceptability, feasibility, sustainability and health-care resources in different country settings.' In 2022 the Ministry of Health of Ethiopia (MoH), will change from MMS to IFA in a set of pilot districts. EPHI and LSHTM have been asked to evaluate the effect of this change on mean birthweight and propose the current trial for this purpose.

The overall aim is to evaluate the programme effectiveness on mean birthweight of providing MMS as part of routine antenatal care, compared to providing IFA.

Findings will support the MoH to make evidence-informed decisions about the large-scale implementation of MMS in Ethiopia and also contribute to the global evidence base on the effectiveness of MMS in a programmatic setting.

Methods: A two-arm cluster randomized trial will be used to estimate the effect of the programme change on mean birthweight, with cost-effectiveness and process evaluations embedded in the trial design.

Women aged 15-49 who deliver a live born child in a study district health facility (mother/infant dyads) will be eligible for enrolment in the study.

The primary outcome measure will be birthweight, recorded in facilities at the time of birth as part of the routine maternity care.

Secondary objectives include costs of providing MMS, acceptability of MMS, adherence to antenatal micronutrient supplementation and implementation challenges.

DETAILED DESCRIPTION:
AIM: The overall aim of the MMS evaluation is to evaluate the programme effectiveness on birthweight of providing MMS as part of routine antenatal care, relative to providing IFA.

STUDY DESIGN: This program effectiveness study involves a cluster randomized trial to estimate the effect of MMS on the primary outcome, birthweight, with embedded cost and process evaluations to measure the secondary objectives.

The overall study design is built around a two-arm, facility-based, cluster randomized trial with district as the unit of randomization (the cluster), whereby districts are randomized to a comparison arm that continues to deliver iron-folic acid supplementation (IFA) as part of the standard antenatal care package, or to an intervention arm where IFA is removed from the standard antenatal care package and replaced with multi-micronutrient supplementation (MMS).

STUDY PERIOD: The entire MMS evaluation will continue for 42 months, starting in March 2022. During 2022, permissions will be obtained and protocols written. In January 2023, a system will be implemented for continuous recording of birth weights in all enrolled health facilities, running until end December 2024 (ie for 24 months). A facility survey will be implemented to collect process data for the secondary objectives at baseline (January 2023), midline (February 2024) and endline (February 2025). Data on costs will be collected alongside the midline facility survey. Primary analysis will be conducted during April 2025.

LOCATION: The evaluation will be done in 42 districts in five regions of Ethiopia. The districts were selected by the Ethiopian Ministry of Health as a pilot area to implement the switch from MMS to IFA as part of routine care, with the intention of also permitting the RCT evaluation of that switch.

42 Districts in detail: Gambella Region (2 districts): Itang especial woreda; Godere;

Somali Region (4 districts): Kebribaya; Ararso; Awbare; Aware;

Oromia Region (20 districts): Gursum; Deder; Goba Koricha; Bele Gesgar; Rayitu; Dodola; Wondo; Kersa; Ejere; Gimbichu; Gemechis; Adami Tulu Jido; Sire; Guna; Medawelabu; Dire; Arero; Becho; Jimma Arjo; Ejersa Lafoo;

Southern Nations Nationalities, and People's Region (12 districts): Sodo; Enemor; Shahsego; Chencha Zuria; Atote Ulo; South Ari; Duguna Fango; Kachabira Bira; Silti; Wonago; Zala; Karat Zuria;

Sidama Region (4 districts): Shebedino; Dara; Aleta chuko; Bona Zuria;

PRIMARY OBJECTIVE: The primary objective is to estimate the effect of MMS implementation on the mean birthweight of babies born in government health facilities to women living in areas where MMS is implemented, relative to the mean birthweight of babies born in government health facilities to women living in areas where standard antenatal IFA supplementation is implemented.

PRIMARY OUTCOME: Birthweight measured as part of routine maternity care will be collected for all live births in enrolled health facilities in intervention and comparison areas.

The protocol for recording the primary outcome, birthweight, will align with routine practices in health facility maternity wards whereby midwives routinely document birthweight. Digital scales will be provided to facilities for this purpose, replacing manual scales. The study team will work with midwives to ensure training in appropriate use of digital scales, accurate recording of birthweight in grammes to four digits, and continuous quality control measures including scale calibration.

SECONDARY OBJECTIVES:

* To estimate the cost and cost-effectiveness of the MMS intervention
* To investigate the processes of MMS implementation including addressing questions about how delivery is achieved and what is actually delivered (fidelity, dose, adaptations, reach and context) and the mechanisms of impact (how providers and clients respond to MMS and any unanticipated pathways or consequences)
* To assess the acceptability and adherence of MMS

SECONDARY ANALYSES AND OBJECTIVES: During the baseline, midline and endline facility surveys data collection tools include: (i) a structured tool to capture detailed information about the antenatal care received by women; (ii) a structured tool to collect data on costs of implementing MMS or IFA; (iii) a structured facility readiness assessment to collect data on availability of services, supplies and trained staff (iv) semi-structured interviews with facility staff on their experience of providing antenatal care services.

The need for additional qualitative interviews with health care users and health care providers to explore emerging topics regarding adherence and acceptability will be reviewed together with the implementation team when implementation has begun and after analysis of baseline data collection.

STUDY POPULATION: For the primary outcome, the study population are mother/infant dyads who are resident in study districts and who access childbirth care in the health centres of those districts. For the secondary objectives there are two study populations: (i) the health staff providing antenatal care services in health centres and (ii) women accessing antenatal care there.

ELIGIBILITY:
Inclusion Criteria:

* For the primary outcome, mothers who deliver a liveborn child in enrolled health facilities and who are willing/consent to participate in the study.
* For the secondary objectives, all antenatal care staff and women attending for routine antenatal care during the survey periods will be included.

Exclusion Criteria:

* For the primary outcome, stillbirths will be excluded. Data for any newborn who subsequently dies while still in the facility will be excluded from all secondary analyses.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population for measurement of birth weight are mother and infant pairs: live newborns born to women who attend enrolled health facilities for childbirth care during the study period in the 42 study districts (clusters). Enrolled health facilities are all government health facilities providing childbirth services that, on average, manage at least 15 births per month (determined by the government database the "District Health Information System"). While acknowledging health-related exclusion criteria, all women attending health facilities for childbirth care in the intervention and comparison districts are potentially eligible for inclusion, irrespective of their place of usual residence or individual characteristics.
Sampling Method: Probability Sample
Enrollment: 25620 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Birthweight | Birthweight from all live births occurring in enrolled facilities between Jan 23 - Dec 24
  The primary objective is to estimate the effect of MMS implementation on the mean birthweight of babies born in government health facilities to women living in areas where MMS is implemented, relative to the mean birthweight of babies born in government health facilities to women living in areas where standard antenatal IFA supplementation is implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Marchant, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Masresha Tessema, PhD, Study Director — Ethiopian Public Health Institute
Locations (6):
- Ethiopia (6):
  - Gambella, Ītang, Gambella Region
  - Oromia, Gīmbīcho, Oromiya
  - Sidama, Bona Gena, Sidama Region
  - SNNPR, Dara, Snnpr Region
  - Somali, Āwarē, Somali
  - Ethiopia Public Health Institute, Addis Ababa

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised data will be made open access using the institutional repository.
  Open access IPD will have no identifiers beyond the study arm allocation and region.
  Data points included will be parity, use of antenatal care services, experience of service use, and birthweight (women) and provision of antenatal care services (health workers).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made open access one year after completion of the primary analysis.
Access Criteria: Full open access to this fully anonymised data.

REFERENCES:
- [Derived] Marchant T, Alemayehu S, Asfaw E, Daba AK, Defar A, Opondo C, Persson LA, Schellenberg J, Taye G, Tesfa A, Tessema B, Zenebe K, Tessema M. Effect of prenatal multiple micronutrient supplementation on birth weight in Ethiopia: protocol for a pragmatic cluster-randomised trial. BMJ Open. 2025 Feb 6;15(2):e093385. doi: 10.1136/bmjopen-2024-093385. PMID 39915025
- [Derived] Berhanu AT, Defar A, Taye G, Daba AK, Alemayehu S, Tessema B, Zenebe K, Opondo C, Tollera G, Hailu M, Schellenberg J, Persson LA, Marchant T, Tessema M. Piloting Multiple Micronutrient Supplementation Within the Routine Antenatal Care System in Ethiopia: Insights From Stakeholders. Matern Child Nutr. 2025 Apr;21(2):e13809. doi: 10.1111/mcn.13809. Epub 2025 Jan 31. PMID 39887615

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT05708183/SAP_000.pdf